CLINICAL TRIAL: NCT05659550
Title: Move With Air: Can a Fan Reduce Exertional Breathlessness During a 4-minute Constant Rate Walking Test in Adults With Cardiopulmonary Disease?
Brief Title: Move With Air: Physiological Response Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dennis Jensen, Ph.D., Associate Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FanEx_2023-9286
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease; Heart Failure
Keywords: Breathlessness; Dyspnea; Exercise; Fan-to-face therapy; Physiological Mechanisms; Constant work rate exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Heart Failure; Dyspnea; Motor Activity

STUDY DESIGN:
Intervention Model Description: Each participant will complete the same constant work rate exercise test under three random-order experiemental conditions.
Masking Description: It is impossible to mask the participants or the investigator since they will be aware if the fan is pointed to the face, to the leg, or there is no fan. However, participants will not be informed of which interventional arm is suspected to be beneficial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fan-to-face (Experimental): The participants will complete a 4-minute constant work rate treadmill test with a basic, portable fan placed in front of the face. The fan will be placed at a location to target the second and third branches of the trigeminal nerve and will be placed a distance chosen by the participant so that the airflow speed is comfortable.
  Interventions: Device: Honeywell HT-900 Turbo Force Air Circulator
- Fan-to-leg (Sham Comparator): The participants will complete a 4-minute constant work rate treadmill test with a basic, portable fan placed in front of the face. The fan will be placed at a location to target the second and third branches of the trigeminal nerve and will be placed a distance chosen by the participant so that the airflow speed is comfortable.
  Interventions: Device: Honeywell HT-900 Turbo Force Air Circulator
- No fan (No Intervention): The participants will complete a 4-minute constant work rate treadmill test with no fan.

INTERVENTIONS:
Device: Honeywell HT-900 Turbo Force Air Circulator — This is a basic, portable, household fan with a single cost of CDN$21.99.
  Other Names: Fan
  Arms: Fan-to-face; Fan-to-leg

SUMMARY:
A fan blowing cool air to the face has been shown to alleviate breathlessness in malignant and non-malignant disease at rest and during exercise, however the underlying physiological mechanisms remain unknown. This random order, three-condition design study will explore physiological mechanisms of breathlessness relief with fan-to-face therapy during constant-rate exercise in people with cardiorespiratory disease.

DETAILED DESCRIPTION:
Constant work rate tests are viewed as the most suitable and sensitive method to assess exertional breathlessness. The 4-minute constant rate treadmill test (4-min CRTT) is a validated test wherein participants exercise at an intensity determined by an incremental test. For the purpose of this study, participants will perform three 4-min CRTT under three random-order experimental conditions: (i) fan to the face; (ii) fan to the leg; (iii) no fan. The intensity of the 4-min CRTTs will be determined based on an exercise endurance test completed in a prior visit: (i) if participants have an endurance time of <3 minutes, they will do each 4-minute CRTT at 50% of peak power output (PPO) achieved on the incremental exercise test, with a fixed grade incline of 40-50% with the speed adjusted to reach 50% PPO; (ii) if participants have an exercise endurance time of 3-8 minutes, they will do each 4-minute CRTT at 75% of peak power output (PPO) achieved on the incremental exercise test, with a fixed grade incline of 60% with the speed adjusted to reach 75% PPO; (iii) if participants have an endurance time of >8 minutes, they will do each 4-minute CRTT at 90% of peak power output (PPO) achieved on the incremental exercise test, with a fixed grade incline of 70-80% with the speed adjusted to reach 90% PPO. This model is based on a recent study on selection of exercise endurance intensities in COPD.Cardiac and dynamic respiratory parameters will be collected breath-by-breath at rest and during exercise using the Hexokin Smart Shirt. In order to target the intranasal pathway located on the trigeminal nerve that is hypothesized to modulate the mechanisms governing the potential effectiveness of a fan to the face, a metabolic cart will be omitted due to the use of the facemask or mouthpiece and nasal clip that would block this pathway.

Using the Borg 0-10 scale, rating of perceived exertion, perceptions of breathlessness intensity, unpleasantness and leg fatigue will be assessed at rest, within the last 15-seconds of each minute of exercise, and at end exercise or the symptom limited peak of exercise. Two areas of facial skin temperature, one at the forehead to target the ophthalmic branch of the trigeminal nerve and the other at the cheek to target the maxillary branch of the trigeminal nerve, will be measured prior to exercise, within the last 15-seconds of each minute of exercise, at end exercise, and following exercise using a medical grade non-contact infrared forehead thermometer. The model number of the forehead thermometer that will be used is THERMOPROPCV2 and is licensed by Health Canada and approved by the U.S. Food and Drug Administration (FDA), CE approved with European health, safety, and environmental protection standards, and approved by the Restriction of Hazardous Substances Directive (RoHS).

ELIGIBILITY:
Inclusion Criteria:

* have a physician diagnosis of cardiopulmonary disease (e.g., chronic obstructive pulmonary disease, interstitial lung disease, heart failure)
* have a body mass index of >18.5 kg/m2 and <35 kg/m2
* must be cleared by a physician to perform physical activity/exercise following the completion of the 'Medical Clearance Form for Cardiopulmonary Exercise Testing'.

Exclusion Criteria:

* have changed their respiratory or cardiac medication dosage and/or frequency of administration in preceding two weeks
* have had a disease exacerbation/hospitalization in preceding six weeks
* have important contraindication(s) to exercise (e.g., significant musculoskeletal or neurological disease) or pulmonary function testing (e.g., eye, chest or stomach surgery, or any history of coughing up significant amounts of blood in the previous 3 months).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Borg modified 0-10 category ratio scale for breathlessness intensity | End-exercise of the 4-minute constant rate treadmill test
  Borg modified 0-10 category ratio scale will be used to assess breathlessness intensity at end-exercise of each 4-minute constant rate treadmill test under three conditions: (i) fan to the face; (ii) fan to the leg (sham) and; (iii) no fan (control). A higher score is indicative of greater breathlessness, while a lower score is indicative of lesser breathlessness.

SECONDARY OUTCOMES:
Cardiopulmonary exercise test (4-minute constant rate) physiological response (ventilatory) | Averaged across the 4-minute constant rate treadmill test
  Mean ventilation (Liters/minute) will be compared across the 4-minute constant rate treadmill tests under the three different conditions: (i) fan to the face; (ii) fan to the leg (sham) and; (iii) no fan (control). A greater mean ventilation is indicative of a less efficient respiratory system, whereas a lower mean ventilation is indicative of a more efficient respiratory system.
Cardiopulmonary exercise test (4-minute constant rate) physiological response (operating lung volumes) | 4 serial dynamic inspiratory capacity maneuvers for each minute of the 4-minute constant rate treadmill test.
  Mean operating lung volumes (i.e., inspiratory capacity in liters) will be compared across the 4-minute constant rate treadmill tests under the three different conditions: (i) fan to the face; (ii) fan to the leg (sham) and; (iii) no fan (control). A greater operating lung volume (i.e., greater inspiratory capacity) is indicative of a better and more efficient breathing pattern, while a lower operating lung volume (i.e., smaller inspiratory capacity) is indicative of a worse and less efficient breathing pattern.
Cardiopulmonary exercise test (4-minute constant rate) physiological response (heart rate) | Averaged across the 4-minute constant rate treadmill test
  Mean heart rate (beats per minute) will be compared across the 4-minute constant rate treadmill tests under the three different conditions: (i) fan to the face; (ii) fan to the leg (sham) and; (iii) no fan (control). A lower heart rate is indicative of better cardiovascular fitness, while a higher heart rate is indicative of worse cardiovascular fitness.
Cardiopulmonary exercise test (3-minute constant rate) physiological response (oxygen saturation) | Averaged across the 4-minute constant rate treadmill test
  Mean oxygen saturation (in percentage) will be compared across the 4-minute constant rate treadmill tests under the three different conditions: (i) fan to the face; (ii) fan to the leg (sham) and; (iii) no fan (control). A lower oxygen saturation is indicative of worse health status, while a higher oxygen saturation is indicative of better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, PhD, Principal Investigator — McGill University
Locations (1):
- Centre of Innovative Medicine of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to Dr. Dennis Jensen's Clinical Exercise and Respiratory Physiology Laboratory page — https://www.mcgill.ca/cerpl/